CLINICAL TRIAL: NCT05167968
Title: Adherence Assesment for Diuretics in Patients Suffering From Precapillary Pulmonary Hypertension
Brief Title: Adherence of Diuretics in Pulmonary Hypertension
Acronym: PHARE
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-A02137-34
Record Dates: First submitted 2021-11-26; First posted 2021-12-22 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Precapillary Pulmonary Hypertension
Keywords: Pulmonary hypertension; Right heart failure; Adherence diuretics
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No intervention (Observational cohort) — For each patient, evaluation and adhesion to diuretics at inclusion are recorded:
  * Self-questioning of medication adherence: Girerd questionnaire
  * Assessment of the Medication Possession Ratio
  * Social and demographic data
  * Comorbidities
  * PH characteristics

SUMMARY:
In this prospective study, the investigators will implement a systematic assessment of adherence to diuretics in a cohort of patients with precapillary pulmonary hypertension.

This study is designed to:

* determine the overall adherence rates for diuretic regimen
* determine the determinants of non-adherence to diuretics
* assess the risk of PH worsening occurrence in the non-adhesion group

DETAILED DESCRIPTION:
Introduction Precapillary pulmonary hypertension (PH) is characterized by remodeling of small pulmonary arteries leading to a progressive increase in pulmonary vascular resistance (PVR) resulting to right heart failure and ultimately death. The prognosis of PH is closely related to the ability of the right ventricle to adapt to the progressive increase in PVR. The occurrence of acute right ventricular decompensation is associated with a very poor prognosis at short term.

The management of precapillary PH is based on specific therapies combined with general measures and supportive therapies. Diuretic treatment is recommended in PAH patients with signs of RV failure and fluid retention (recommendation class I, level of evidence C). The beneficial effect of diuretics is probably essential for preventing episodes of acute right ventricular decompensation. However, no study analyzed the rate of adherence to diuretic regimen in PH patients and the impact of patterns of adherence to diuretics on the outcomes of patients.

Aim and objectives

The main objectives of this study are to:

* determine the overall adherence rates for diuretic regimen
* determine the determinants of non-adherence to diuretics
* assess the risk of PH worsening occurrence in the non-adherence group

Methodology

Evaluation of subjects and adhesion to diuretics at inclusion are recorded:

* Self-questioning of medication adherence: Girerd questionnaire
* Assessment of the Medication Possession Ratio
* Social and demographic data
* Comorbidities
* PH characteristics
* Clinical evaluation: dyspnea assessed by NYHA functional class (New York Heart Association Functional Classification : I-IV), signs of right heart failure
* Type of treatment regimen
* History of serious events including non-programmed hospitalization for PH and/or worsening of the disease (15% reduction in the 6-minute walking test and worsening of the WHO functional class) and/or the need to reinforce specific PH therapies

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old
* Precapillary PH
* Diuretics treatment for at least 12 months
* Having given his/her non-opposition to participate

Exclusion Criteria:

* Treatment regimen without diuretics
* Diuretics treatment for less than 12 months
* Postcapillary PH
* People refusing or unable to give informed consent
* No affiliation to a regime of social security.
* Protected patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with Precapillary PH and diuretics treatment for at least 12 months, at least 18 years old
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2022-01-13 (Actual); Primary Completion 2024-01-24 (Actual); Study Completion 2024-01-24 (Actual)

PRIMARY OUTCOMES:
Score of Girerd (French self-administered questionnaire about adherence medication) and level of medication possession ratio (MPR) | 2 weeks previous hospitalization
  Prevalence of high adherence to diuretics in PH patients
  Girerd questionnaire is made up of 6 items which are evaluated in a binary way : Yes = 0 point & No = 1 point. Three medication categories are defined : high adherence (score = 6), moderate adherence (score = 4 or 5) and low adherence (score < or = 3). MPR is defined by the ratio between the number of days during which the patient is supplied for his medication and the number of days during he should be supplied his medication, over a given period (12 months). Patients with a MPR > 0,80 are considered to have a high adherence whereas patients with a MPR < 0,80 are considered to have a low adherence to diuretics.

SECONDARY OUTCOMES:
To determine the determinants of non-adherence to diuretics | 30 months previous hospitalization
  Determinants related to the patient, treatment, disease and care will be recorded.
  Association between selected determinants and adherence to diuretics will be analyzed
To assess the risk of PH worsening occurrence in the non-adhesion group | 30 months previous hospitalization
  Occurrence of serious events including non-programmed hospitalization for PH and/or worsening of the disease (15% reduction in the 6-minute walking test and worsening of the WHO functional class) and/or the need to reinforce specific within the 12 months preceding inclusion.
  Comparison of serious event prevalence in the high- and low-adherence groups

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Camille Chaumais, PharmD, PhD, Principal Investigator — Bicêtre Hospital
Locations (1):
- Hospital Bicêtre - Pneumology department, Le Kremlin-Bicêtre, France

IPD SHARING:
Plan to Share IPD: No